CLINICAL TRIAL: NCT05465265
Title: Pre-Exposure Prophylaxis for Prevention of Human Immunodeficiency Virus Transmission Among Sexual and Injecting Partners of People Who Inject Drugs in Nairobi, Kenya
Brief Title: PrEP for Prevention of HIV Transmission Among People Who Inject Drugs in Nairobi, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenyatta National Hospital (Other Government); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Cosmas Gitobu, Principal investigator as a Post doctoral fellowship candidate, University of Washington, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00013701; 3D43TW009345-10S6 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: HIV Antibody Positivity; PrEP Uptake
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: The study may have two arms: "Cases will be navigated into PrEP services" and the "Control group will just be given PrEP information pamphlets"
Who Masked: Care Provider
Masking Description: Cases : Navigation into PrEP
  Control group: Provision of pamphlets with information on PrEP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention and control group (Active Comparator): To establish the effect of navigation on PrEP uptake, adherence and retention among PWID.
  Interventions: Behavioral: Navigation into prEP by use of PrEP-UP intervention (provision of PrEP information through 5 counselling sessions, peer support, booking of appointments for PWIDs)
- Control group (Placebo Comparator): To establish the effect of providing PrEP information through pamphlets on PrEP uptake, adherence and retention among PWID.
  Interventions: Behavioral: Navigation into prEP by use of PrEP-UP intervention (provision of PrEP information through 5 counselling sessions, peer support, booking of appointments for PWIDs)

INTERVENTIONS:
Behavioral: Navigation into prEP by use of PrEP-UP intervention (provision of PrEP information through 5 counselling sessions, peer support, booking of appointments for PWIDs) — Cases: Navigation of PWID into PrEP-Navigation into prEP by use of PrEP-UP intervention (provision of PrEP information through 5 counselling sessions, peer support, booking of appointments for PWIDs) Control group: Provision of PrEP information to PWID through pamphlets on PrEP uptake, adherence and retention among PWID.
  Other Names: Control Group: Provision of PrEP pamphlets has is expected to have no effect on uptake of PrEP, adherence to PrEP and retention into PrEP

SUMMARY:
The investigators broadly aim at determining barriers and facilitators to PrEP uptake and adherence and retention among the study participants. The investigators have the following specific objectives of determining: (1) the PrEP knowledge levels, attitudes, practices, and user experiences among injecting and sexual partners of PWID in Nairobi County (2) the socio-demographic, behavioural, and structural factors hindering the uptake of PrEP among PWID's sexual and injecting partners in Nairobi County; and (3) the effect of a theory-guided behavioural intervention (PrEP-UP) utilizing peer outreach and navigation on the uptake of PrEP by the study participants.

The investigators hypothesize that: PWID's injecting and sexual partners in Nairobi City lack PrEP knowledge, and have poor attitudes practices, and user experiences about PrEP; less than 50.0% of the PWID's sexual and injecting partners in Nairobi County have socio-demographic, behavioural and structural factors hindering their uptake of PrEP; and a theory-guided behavioural intervention (PrEP-UP) utilizing peer outreach and navigation has no effect on the uptake of PrEP by the study participants.

DETAILED DESCRIPTION:
Background: The annual global number of new HIV infections among adults has remained unchanged over the last decade and it is largely fuelled by key populations among them people who inject drugs (PWID). Key populations in Kenya account for one-third of all new HIV infections and 18.3% of PWID in the country are living with HIV. Drug and substance use is on the increase in the country, with close to 4 out of 10 Kenyans reporting to have used a substance in their lifetime including injectable drugs thus fueling the spread of HIV. Pre-Exposure Prophylaxis (PrEP) is effective in the prevention of HIV transmission among PWID by over 70.0% if and when used correctly. However, uptake, adherence, scale-up of use, coverage and retention currently remain limited. Thus, effective interventions are needed to enhance the uptake of PrEP among PWID and their sexual and injecting partners in order to prevent HIV transmission.

Objectives of the Study: Broadly, the investigators aim at determining PrEP uptake barriers and facilitators and adherence among the study participants and the sequel of a theory-guided behavioral intervention model (PrEP-UP) on the uptake of PrEP by the study participants. Specifically, the investigators aim at determining: (1) the PrEP knowledge levels, attitudes, practices and user experiences among the study participants(2) the socio-demographic, behavioural and structural factors hindering the uptake of PrEP among the study participants; and (3) the effect of a theory-guided behavioural intervention (PrEP-UP) utilizing peer outreach and navigation on the uptake of PrEP by the study participants.

Methods: The investigators will conduct the study for twelve months (1st July 2021 to 30th June 2022) and they will use an implementation study through a pre-post design to assess 256 participants' self-reported PrEP uptake and retention before and after exposure to a theory-guided behavioural intervention (PrEP-UP) utilizing navigators and peer outreach for the 128 'cases' and PrEP information Pamphlet and list of health facilities offering PrEP for free in Nairobi County for the 128 'control' group members. The investigators will use four study sites namely Githurai, Kawangware, Ngara and Pangani PWID's hotspots within Nairobi City. The targeted study participants are PWID's sexual and injecting partners of ages 18 years and above. The investigators will recruit 256 study participants into the study by use of peers and social workers in the University of Washington's Needle and Syringe Program (NSP) sites in Githurai, Kawangware, Ngara and Pangani. The investigators will collect baseline data after recruitment while the interventions for both groups will be offered in a maximum 5 contact sessions with investigators and a follow-up of the participants will be done by the investigators at weeks 4, 8 and 12 to establish whether study participants have taken up PrEP by week 12 during which post-intervention data will be collected. Lastly, participants' self-reported PrEP retention will be documented by investigators at 18 weeks and HIV tests will be conducted on the participants by the investigators (optional) through OraQuick antibody HIV tests. The investigators will analyze: quantitative data through the Statistical Package for Social Sciences (SPSS) version 24 and: qualitative data through flow chart matrices to establish divergence and convergence of themes.

Significance of the Study: Through the study, the investigators will contribute to the global call for the reduction in new HIV infections among PWIDs and their sexual and injecting partners. The study will further inform the investigators on the effectiveness-implementation science interventions and recommend the best PrEP scale-up approaches in addition to contributing to the global scientific knowledge.

ELIGIBILITY:
The inclusion criteria for the study includes:

Being age 18 years and above.

Being HIV negative on a rapid HIV test conducted prior to interviews.

No pregnancy for females at the time of recruitment.

Active injection of illicit drugs in the six months preceding the study.

High multiple HIV risk and high HIV through sexual activities and sharing of injection equipment or syringes (the high multiple-risk group mixed unsafe drug use with unsafe sexual practices; the second group practiced high-risk sex with non-consistent condom combined with drug use; the moderate-risk group had limited unsafe sexual practices; and the "low-risk" group never had unprotected sex and never shared needles and other injection equipment).

Informed consent to participate inti the study.

The exclusion criteria includes:

Being a minor (below 18 years).

Those not actively injecting drugs.

Acute or chronic HIV infection

Those not consenting to participation into the study.

Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
PrEP uptake following either navigation or provision of pamphlets (Self-reported uptake reported through quantitative interviews) | 12 weeks
  Outcome 1: Uptake of PrEP following the study interventions (either navigation into PrEP or pamphlets) Outcome 2-Adherence to PrEP Outcome 3: Retention into PrEP following uptake
Retention into PrEP after uptake following either navigation or provision of pamphlets (Self-reported retention) | 18 weeks
  Retention into PrEP for 18 weeks (self-reported through interviews conducted by investigators))
Adherence to PrEP for 18 weeks (self reported through interviews conducted by investigators) | 18 weeks
  Adherence to PrEP after uptake following either navigation or provision of pamphlets (Self-reported adherence through interviews conducted by investigators)

SECONDARY OUTCOMES:
HIV Status following Rapid HIV tests OraQuick rapid HIV 1 antibody tests | 18 weeks
  Seroconversion following PreP uptake or failure to take up PrEP in the 18 weeks of the RCT

CONTACTS AND LOCATIONS:
Overall Officials: Cosmas Gitobu, Principal Investigator — University of Washington
Locations (1):
- Pangani DIC, Ngara DIC, Githurai DIC, Kawangware DIC, Nairobi, Nairobi County, Kenya